CLINICAL TRIAL: NCT02600715
Title: Reduction of Bladder Injection Pain With Belladonna Opiate Suppository: A Randomized, Double-Blind, Placebo-Controlled Trial (ROBIN Trial)
Brief Title: Reduction of Bladder Injection Pain With Belladonna Opiate Suppository
Acronym: ROBIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Edgar LeClaire, MD (Other)
Responsible Party: Sponsor-Investigator, Edgar LeClaire, MD, Clinical Instructor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00003056; 15-051 (Other: Wichita Medical Research and Education Foundation IRB)
Record Dates: First submitted 2015-10-29; First posted 2015-11-09 (Estimated); Results first posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-06

CONDITIONS: Overactive Bladder; Urinary Urge Incontinence; Urinary Bladder, Neurogenic; Painful Bladder Syndrome
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urinary Bladder, Neurogenic; Cystitis, Interstitial | interventions — Botulinum Toxins, Type A; Idoxuridine; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active B&O suppository of belladonna (Experimental): Receive the B&O suppository (belladonna/morphine) 40 minutes prior to Onabotulinumtoxin A (BoNT) injection procedure in conjunction with local analgesia.
  Interventions: Drug: Onabotulinumtoxin A (BoNT); Drug: belladonna; Drug: Morphine; Drug: Active B&O suppository of belladonna
- Placebo suppository (Placebo Comparator): Receive a placebo suppository 40 minutes prior to Onabotulinumtoxin A (BoNT) injection procedure in conjunction with local analgesia.
  Interventions: Drug: Onabotulinumtoxin A (BoNT); Drug: Placebo

INTERVENTIONS:
Drug: Onabotulinumtoxin A (BoNT)
  Other Names: Botox; Allergan
Drug: belladonna — Part of dosage of the compounded active B&O suppository of belladonna 16.2mg and morphine 7.5mg.
  Arms: Active B&O suppository of belladonna
Drug: Morphine — Part of dosage of the compounded active B&O suppository of belladonna 16.2mg and morphine 7.5mg.
  Arms: Active B&O suppository of belladonna
Drug: Placebo — matching placebo to B&O suppository
  Arms: Placebo suppository
Drug: Active B&O suppository of belladonna — belladonna 16.2mg and morphine 7.5mg
  Arms: Active B&O suppository of belladonna

SUMMARY:
The purpose of this study is to test whether using belladonna & opiate suppositories (B&Os) can improve patient discomfort during Onabotulinumtoxin A (BoNT) injection into the bladder for treatment of overactive bladder, neurogenic detrusor overactivity, or interstitial cystitis.

ELIGIBILITY:
Inclusion Criteria:

* Met clinical criteria under outside care or during the Principal Investigator's routine standard of care for BoNT injection therapy
* No contraindication to BoNT therapy as outlined by drug manufacturer guidelines
* Participants have elected to have the BoNT injection therapy prior to being offered enrollment into the study for either overactive bladder (OAB), neurogenic detrusor overactivity (NDO), or refractory interstitial cystitis (IC)

Exclusion Criteria:

* Currently pregnant
* Currently nursing a baby
* Anticipated geographic relocation within the first 3 months following treatment
* Allergy to morphine, belladonna, or opiates
* Patients will be excluded if participating in another research study
* Individuals unable to provide informed consent or to complete two-week follow-up bladder testing (post-void residual) or data collection will also be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar LeClaire, MD, FACOG, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - Wichita Women's Pelvic Surgery Center at Associates in Women's Health, Wichita, Kansas
  - University of Kansas School of Medicine - Wichita, Wichita, Kansas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began December 1, 2015 at a private urogynecology clinic. There were 32 patients that were assessed for eligibility. Four patients were excluded: three patients did not meet inclusion criteria (did not proceed with in-office treatment) and one patient declined to participate due to wanting the active suppository.
Pre-assignment Details: 28 patients consented to participate in the study. Two patients withdrew consent to participate and did not end up participating: one patient's medication resumed efficacy, and one patient withdrew regarding possible use of narcotics and concern due to a a previous narcotic addition.
  Thus, only 26 patients are considered enrolled in this study.
Groups:
- Active Belladonna & Opiate (B&O) Suppository: Receive the B&O suppository (belladonna/morphine) 40 minutes prior to Onabotulinumtoxin A (BoNT) injection procedure in conjunction with local analgesia.
  Onabotulinumtoxin A (BoNT)
  belladonna: Part of dosage of the compounded active B&O suppository of belladonna 16.2mg and morphine 7.5mg.
  Morphine: Part of dosage of the compounded active B&O suppository of belladonna 16.2mg and morphine 7.5mg.
  Active B&O suppository of belladonna: belladonna 16.2mg and morphine 7.5mg
- Placebo Suppository: Receive a placebo suppository 40 minutes prior to Onabotulinumtoxin A (BoNT) injection procedure in conjunction with local analgesia.
  Onabotulinumtoxin A (BoNT)
  Placebo: matching placebo to B&O suppository
Period: Overall Study
Arm/Group | Active Belladonna & Opiate (B&O) Suppository | Placebo Suppository
Started | 13 | 13
Allocated to Randomization | 13 | 13
Received Treatment and Suppository | 13 | 13
Completed 2-week Follow-up Appointment | 13 | 12
Completed (Included in final analysis) | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active B&O Suppository of Belladonna: Receive the B&O suppository (belladonna/morphine) 40 minutes prior to Onabotulinumtoxin A (BoNT) injection procedure in conjunction with local analgesia.
  Onabotulinumtoxin A (BoNT)
  belladonna: Part of dosage of the compounded active B&O suppository of belladonna 16.2mg and morphine 7.5mg.
  Morphine: Part of dosage of the compounded active B&O suppository of belladonna 16.2mg and morphine 7.5mg.
  Active B&O suppository of belladonna: belladonna 16.2mg and morphine 7.5mg
- Total: Total of all reporting groups
Arm/Group | Active B&O Suppository of Belladonna | Placebo Suppository | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.62 (10.25) | 65.54 (10.22) | 69.58 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 35.45 (11.34) | 34.19 (6.33) | 34.82 (9.02)
Vaginal parity [Median (Inter-Quartile Range); unit: pregnancies] — Vaginal parity is the number of pregnancies that the patient had, that was carried to greater 20 weeks.
  Zero indicates that the patient did not have any pregnancies beyond 20 weeks (nulliparous).
  pregnancies | 2 [2 to 3] | 3 [1 to 3] | 2 [2 to 3]
Current smoker [Count of Participants; unit: Participants] | 1 | 1 | 2
Menopausal [Count of Participants; unit: Participants] | 13 | 12 | 25
Estrogen use [Count of Participants; unit: Participants]
  Vaginal estrogen | 4 | 7 | 11
  Oral estrogen | 2 | 1 | 3
Gynecologic disorders/diagnoses [Count of Participants; unit: Participants]
  Vulvovaginal atrophy | 7 | 7 | 14
  Constipation | 1 | 2 | 3
  Chronic cystitis | 3 | 2 | 5
  Cystocele | 0 | 3 | 3
  Vaginal vault prolapse | 1 | 2 | 3
  Uterine prolapse | 0 | 0 | 0
  Rectocele | 0 | 1 | 1
Medication use [Count of Participants; unit: Participants]
  Steroid medication | 1 | 0 | 1
  Narcotic medication | 1 | 1 | 2
  Diuretic medication | 1 | 4 | 5
Surgical history [Count of Participants; unit: Participants]
  Hysterectomy | 10 | 10 | 20
  Bilateral salpingo-oophorectomy (BSO) | 6 | 7 | 13
  Prolapse surgery with mesh | 0 | 1 | 1
  Prolapse surgery without mesh | 2 | 3 | 5
  Previous sling procedure | 3 | 3 | 6
  Laparotomy | 5 | 5 | 10
  Back or spinal surgery | 3 | 2 | 5
Medication use in Last 24 Hours [Count of Participants; unit: Participants] — Participant medication use in last 24 hours prior to intravesical onabotulinum toxin A injection
  Participants
    Selective serotonin reuptake inhibitors (SSRIs) | 7 | 0 | 7
    Nonsteroidal anti-inflammatory drugs (NSAIDs) | 5 | 6 | 11
    Sedative medication | 1 | 5 | 6
    Neuromodulator medication | 1 | 1 | 2
    Opioid medication | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Bladder Injection Pain
Description: The primary outcome will be calculated difference in numeric rating scale (NRS) pain score prior to procedure and midway through procedure. Scale is one question and has a range from a score of 0 (no pain) to 10 (worst possible pain). Measure will be reported as the intraoperative pain score minus the preoperative pain score.
Time Frame: Baseline and intraoperative
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Total: 26 participants
Arm/Group | Active B&O Suppository of Belladonna | Placebo Suppository | Total
Number analyzed (Participants) | 13 | 13 | 26
units on a scale | 5 [2 to 6] | 4 [3 to 5] | 5 [2 to 6]
Statistical Analysis 1: Comparison: Active B&O Suppository of Belladonna vs Placebo Suppository; Test type: Equivalence — Test for differences in continuous variables; p = 0.94, Kruskal-Wallis — Two-sided alpha of 0.05 was used to determine statistical significance

2. Secondary Outcome: Pre-analgesia Pain Score
Description: Measured using NRS. Scale is one question and has a range from a score of 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active B&O Suppository of Belladonna | Placebo Suppository | Total
Number analyzed (Participants) | 13 | 13 | 26
units on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Post-operative Pain Score
Description: Measured using NRS. Scale is one question and has a range from a score of 0 (no pain) to 10 (worst possible pain).
Time Frame: Postoperative (within 10 minutes of the end of the BoNT procedure)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active B&O Suppository of Belladonna | Placebo Suppository | Total
Number analyzed (Participants) | 13 | 13 | 26
units on a scale | 2 [0 to 5] | 3 [1 to 7] | 2 [1 to 5]

4. Secondary Outcome: Number of Participants Declining to Complete Procedure Due to Pain Intolerance
Description: Number of patients that decline to proceed with entire procedure (20 injections) due to pain or discomfort.
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Active B&O Suppository of Belladonna | Placebo Suppository | Total
Number analyzed (Participants) | 13 | 13 | 26
Participants | 0 | 0 | 0

5. Secondary Outcome: Postoperative Voiding Trial Results
Description: Distribution of patients with postoperative volume in ml of post-void residual urine obtained via catheter greater than 200ml.
Time Frame: Postoperative (before leaving the clinic, within 3 hours of the end of the BoNT procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | Active B&O Suppository of Belladonna | Placebo Suppository | Total
Number analyzed (Participants) | 13 | 13 | 26
Participants | 3 | 5 | 8

6. Secondary Outcome: Post Void Residual (PVR)
Description: Distribution of patients with volume in ml of post-void residual urine obtained via catheter greater than 200 ml at 2-week follow-up appointment.
Time Frame: 2 Weeks
Population: One patient did not complete 2-week follow-up post-void residual exam.
Measure: Count of Participants; unit: Participants
Groups:
- Total: 25 participants
Arm/Group | Active B&O Suppository of Belladonna | Placebo Suppository | Total
Number analyzed (Participants) | 13 | 12 | 25
Participants | 2 | 3 | 5

7. Secondary Outcome: Number of Participants With Evidence of Infection or Positive Urine Culture
Description: Urinalysis results showing evidence of infection or positive urine culture at 2-week follow-up appointment.
Time Frame: 2 Weeks
Population: One patient did not complete 2-week follow-up appointment.
Measure: Count of Participants; unit: Participants
Arm/Group | Active B&O Suppository of Belladonna | Placebo Suppository | Total
Number analyzed (Participants) | 13 | 12 | 25
Participants | 2 | 4 | 6

8. Secondary Outcome: Participant Satisfaction With Pain Control
Description: Measured using one question Likert scale. This will be a 4-level scale ranging from 'not at all satisfied,' 'slightly satisfied,' 'mostly satisfied,' and 'very much satisfied.'
Time Frame: Postoperative (within 10 minutes of the end of the BoNT procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | Active B&O Suppository of Belladonna | Placebo Suppository | Total
Number analyzed (Participants) | 13 | 13 | 26
Participants
  Not at all satisfied | 0 | 1 | 1
  Slightly satisfied | 2 | 1 | 3
  Mostly satisfied | 2 | 5 | 7
  Very much satisfied | 9 | 6 | 15

ADVERSE EVENTS:
Time Frame: Two-weeks
Description: Adverse event reporting is applicable to only participants that completed the two week follow-up visit post-operative. Thus, only 25 participants are included.
Groups:
- Total: 25 participants completed the two-week follow-up visit
Arm/Group | Active B&O Suppository of Belladonna | Placebo Suppository | Total
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/25
Other Adverse Events (participants affected / at risk) | 2/13 | 4/12 | 6/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active B&O Suppository of Belladonna (N=13) | Placebo Suppository (N=12) | Total (N=25)
Urinary Tract Infection Two Weeks Post-operative (Infections and infestations) | 2 (13) | 4 (12) | 6 (25) — At the two week follow-up appointment, when indicated, specimens were sent for confirmatory culture if urinalysis indicated infection and empiric antibiotic treatment was initiated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-11-05): https://cdn.clinicaltrials.gov/large-docs/15/NCT02600715/Prot_SAP_000.pdf
  • Informed Consent Form (2015-11-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT02600715/ICF_001.pdf